CLINICAL TRIAL: NCT00110006
Title: Prognostic Significance of Early Positron Emission Tomography (PET) With Fluorine-18 Fluorodeoxyglucose ([18F] FDG) in Intermediate and High Grade Non-Hodgkin's Lymphoma
Brief Title: Positron Emission Tomography Using Fludeoxyglucose F 18 in Predicting Response to Treatment in Patients Who Are Receiving Rituximab and Combination Chemotherapy for Newly Diagnosed Non-Hodgkin's Lymphoma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No accrual
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Panayiotis Savvides, MD, Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CASE2404; P30CA043703 (NIH); CASE-CWRU-2404 (Other: Case Comprehensive Cancer Center); CWRU-100401
Record Dates: First submitted 2005-05-03; First posted 2005-05-04 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-06

CONDITIONS: Lymphoma
Keywords: contiguous stage II grade 3 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; stage I grade 3 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 3 follicular lymphoma; contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; stage I adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma; contiguous stage II mantle cell lymphoma; noncontiguous stage II mantle cell lymphoma; stage I mantle cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; anaplastic large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell; Lymphoma, Large-Cell, Anaplastic | interventions — Rituximab; Cyclophosphamide; Doxorubicin; Prednisone; Vincristine; Magnetic Resonance Spectroscopy; Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: rituximab — Rituximab IV over 3-6 hours. Treatment repeats every 14-21 days for up to 4 courses in the absence of unacceptable toxicity.
Drug: cyclophosphamide — Cyclophosphamide IV over 30 minutes. Treatment repeats every 14-21 days for up to 4 courses in the absence of unacceptable toxicity.
Drug: doxorubicin hydrochloride — Doxorubicin IV over 5 minutes. Treatment repeats every 14-21 days for up to 4 courses in the absence of unacceptable toxicity.
Drug: prednisone — Oral prednisone once daily on days 1-5. Treatment repeats every 14-21 days for up to 4 courses in the absence of unacceptable toxicity.
Drug: vincristine sulfate — Vincristine IV over 5 minutes on day 1. Treatment repeats every 14-21 days for up to 4 courses in the absence of unacceptable toxicity.
Procedure: positron emission tomography — Beginning 1 hour after receiving fludeoxyglucose F 18, patients undergo whole-body positron emission tomography (PET) scanning. Patients undergo repeat ^18FDG-PET scanning between days 7-10 of course 1, between courses 3 and 4, and then at the completion of R-CHOP.
Radiation: fludeoxyglucose F 18 — Patients receive fludeoxyglucose F 18 (^18FDG) IV.

SUMMARY:
RATIONALE: Diagnostic procedures, such as positron emission tomography (PET) using fludeoxyglucose F 18, may help in learning how well chemotherapy works to kill cancer cells and allow doctors to plan better treatment. Comparing results of diagnostic procedures done before, during, and after chemotherapy may help doctors predict a patient's response to treatment and help plan the best treatment.

PURPOSE: This clinical trial is studying positron emission tomography using fludeoxyglucose F 18 to see how well it works in predicting response to treatment in patients who are receiving rituximab and combination chemotherapy for newly diagnosed non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the positive and negative predictive values of early positron emission tomography (PET) scanning using fludeoxyglucose F 18 in terms of the probability of patients with newly diagnosed intermediate- or high-grade non-Hodgkin's lymphoma who achieve or do not achieve complete remission, after treatment with 1 course of rituximab and combination chemotherapy comprising cyclophosphamide, doxorubicin, vincristine, and prednisone.
* Determine event free and overall survival of patients with an early positive and negative PET scan treated with this regimen.
* Determine the predictive value of early PET scan response ratio as a continuous variable in terms of response to therapy (assessed at the end of therapy), disease-free survival, and overall survival, in patients treated with this regimen.
* Correlate International Prognostic Index score at presentation with early PET scan results and overall outcome in patients treated with this regimen.
* Correlate the degree of neutropenia 7 to 10 days after the first course of treatment with rituximab and combination chemotherapy with PET scan response and pre-treatment blood CD34-positive cell concentration in these patients.

OUTLINE: This is a multicenter study.

Patients receive fludeoxyglucose F 18 (^18FDG) IV. Beginning 1 hour later, patients undergo whole-body positron emission tomography (PET) scanning. Patients also undergo conventional radiographic staging of their disease.

Patients then receive standard R-CHOP (or an alternative regimen) comprising rituximab IV over 3-6 hours, cyclophosphamide IV over 30 minutes, doxorubicin IV over 5 minutes, and vincristine IV over 5 minutes on day 1 and oral prednisone once daily on days 1-5. Treatment repeats every 14-21 days for up to 4 courses in the absence of unacceptable toxicity.

Patients undergo repeat ^18FDG-PET scanning between days 7-10 of course 1, between courses 3 and 4, and then at the completion of R-CHOP. Patients also undergo radiographic restaging of their disease between courses 3 and 4 and at the completion of R-CHOP.

After completion of study treatment, patients are followed every 3-4 months for 2 years, every 6 months for 1 year, and then annually for 3 years.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed newly diagnosed non-Hodgkin's lymphoma (NHL)

  * Intermediate- or high-grade disease
  * Stage I-IV disease
  * Any of the following subtypes are allowed:

    * Diffuse large B-cell lymphoma
    * Anaplastic large cell lymphoma
    * Mantle cell lymphoma
    * Grade 3 follicular lymphoma
    * Mediastinal B-cell lymphoma
  * The following subtypes are not allowed:

    * Lymphoblastic lymphoma
    * Mycosis fungoides/Sézary's syndrome
    * HTLV-1 associated T-cell leukemia or lymphoma
    * Primary CNS lymphoma
    * HIV-associated lymphoma
    * Transformed lymphoma
    * Burkitt's lymphoma
* Adequate staging of lymphoma by any of the following methods:

  * CT scan or MRI of affected sites
  * Unilateral or bilateral bone marrow biopsy
  * Positive pre-treatment positron emission tomography (PET) scan
  * Lumbar puncture
* Radiographically measurable disease by PET scan
* Any International Prognostic Index risk category allowed
* No prior diagnosis of another hematologic malignancy NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count > 1,000/mm^3*
* Platelet count ≥ 75,000/mm^3* NOTE: *Unless due to NHL

Hepatic

* Bilirubin ≤ 2.0 mg/dL* (excluding Gilbert's disease) NOTE: *Unless due to NHL

Renal

* Creatinine ≤ 2.0 mg/dL (unless due to NHL)

Cardiovascular

* Ejection fraction ≥ 45% by echocardiogram or MUGA

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No other malignancy within the past 5 years except superficial nonmelanoma skin cancer or carcinoma in situ of the cervix
* No other serious co-morbid disease that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior rituximab for NHL
* No concurrent filgrastim [G-CSF] during course 1 of study treatment except for patients > 70 years of age OR patients with active infection

Chemotherapy

* No prior chemotherapy for NHL

Endocrine therapy

* No prior steroids for NHL

Radiotherapy

* No prior radiotherapy for NHL
* Concurrent consolidation radiotherapy to sites of bulky disease allowed at the discretion of the attending physician

Surgery

* Not specified

Other

* No other prior treatment for NHL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2004-12

PRIMARY OUTCOMES:
Complete remission as measured by positron emission tomography (PET) at 7-10 days after R-CHOP, and after completion of study treatment | at 7-10 days after R-CHOP, and after completion of study treatment
Overall survival at 7-10 days after R-CHOP, and after completion of study treatment | at 7-10 days after R-CHOP, and after completion of study treatment
Disease-free survival at 7-10 days after R-CHOP, and after completion of study treatment | at 7-10 days after R-CHOP, and after completion of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Panayiotis Savvides, MD, Study Chair — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center